CLINICAL TRIAL: NCT03843073
Title: Evaluation of the Safety and Clinical Performance of the Gen 2 Connected Catheter - Wireless Urinary Prosthesis for Management of Chronic Urinary Retention
Brief Title: Connected Catheter- Safety and Effectiveness Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigation of this device has been transitioned into a new study by the sponsor. The data generated in this study will not be used to support a marketing application
Sponsor: Spinal Singularity (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CIP-0001 (Formerly ES-01)
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Urinary Retention; Neurogenic Bladder; Urologic Diseases
Keywords: Spinal Cord Injury (SCI),; Neurogenic Lower Urinary Tract Dysfunction (NLUTD); Catheter associated Urinary Tract Infection (CAUTI); Urinary Catheters; Urinary Retention; Enlarged Prostate; Prostate cancer
MeSH Terms: conditions — Urinary Retention; Urinary Bladder, Neurogenic; Urologic Diseases; Spinal Cord Injuries; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Connected Catheter Users (Experimental)
  Interventions: Device: Connected Urinary Catheter

INTERVENTIONS:
Device: Connected Urinary Catheter — Patients will use the Connected Catheter to empty the bladder during the course of treatment.

SUMMARY:
The Connected Catheter is a fully internal, urethral indwelling urinary prosthesis designed for improved bladder management in males with urinary retention disorders requiring catheterization. It is a sterile, extended-use device that resides fully internally to the male lower urinary tract for an intended use life of up to 7 days per catheter.

DETAILED DESCRIPTION:
Spinal Singularity has developed the Connected Catheter System to address several drawbacks of urinary catheters. The Connected Catheter is fully internal, indwelling urinary prosthesis designed for improved bladder management in males with urinary retention disorders requiring catheterization. Each subject will use the Connected Catheter for up to 35-40 days. This includes five device exchange appointments. The appointments are spaced 7 days apart and at each appointment the catheter will be replaced with a new one. Additionally, weekly follow-up will occur for 14 days following the final appointment after the subject discontinues use of study device and reverts to his original catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Males age ≥ 18 with clinical diagnosis of significant urinary retention
2. Must be clinically suitable and capable of safely managing bladder using an intermittent voiding or indwelling strategy

   Must have stable urinary management history as determined by the Investigator

   OR:

   Must have urodynamic profile suitable for the Gen 2 Connected Catheter (including bladder capacity > 200mL without uninhibited bladder contractions)
3. Subject's lower urinary tract anatomy must fall within the ranges serviceable by the Gen 2 Connected Catheter device, as specified in the Investigational Device Instructions for use (IFU)

Exclusion Criteria:

1. Active symptomatic urinary tract infection (UTI), as defined in this protocol (subjects may receive the device after UTI has been treated)
2. Significant risk profile or recent history of urethral stricture (e.g. stricture within past 90 days)
3. Significant risk profile or recent history of clinically significant (uncontrolled) autonomic dysreflexia (AD)
4. Significant intermittent urinary incontinence (between catheterizations)
5. Uninhibited bladder contractions and/or Vesicoureteral reflux that is not reliably controlled with medication or alternate therapy (e.g. Botox injections)
6. Pre-existing urinary pathologies and/or morphological abnormalities of the lower urinary tract or bladder (assessed during in-depth medical screening, including cystoscopy and urine analysis)

   1. Urinary tract inflammation or neoplasm
   2. Urinary fistula
   3. Bladder diverticulum (outpouching) > 5cm in size
   4. Chronic pyelonephritis (secondary to upper urinary tract infection(s) within past 6 months)
   5. Impaired kidney function or renal failure
   6. Active gross hematuria
   7. Active urethritis
   8. Bladder stones
7. Dependence on an electro-magnetic medical implant (e.g. cardiac pacemaker or implanted drug pump) or external device
8. Any unsuitable comorbidities as determined by the investigator or complications related to use of certain medications
9. Any physical or cognitive impairments that diminish the subject's ability to follow directions or otherwise safely use the Connected Catheter System
10. Catheter Assessment Tool screening yields unacceptable results

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Successful Bladder Emptying Using Connected Catheter | 35-40 days
  Rate of participants with successful voiding using the Connected Catheter as assessed by Post-Residual Volume (PVR) measurement via ultrasound
  A subject is considered a responder to the treatment if a minimum of 80% of their PVR values met the following criteria
  PVR is ≤ 50 mL OR PVR is ≤ baseline PVR with the standard of care catheter
Rate of device related Serious Adverse Events | 0 - 40 days
  Rate of participants treated with the Connected Catheter reported with a serious device related adverse event

SECONDARY OUTCOMES:
Successful device insertion, anchoring, and removal | 35-40 days
  Rate of Connected Catheter successfully inserted, anchored and removed
Successful sealing of the catheter valve | 35-40 days
  Rate of Connected Catheter valves sealed successfully
Quality of life improvement as measured by SCI-QOL Survey and other surveys | 35-40 days
  Rate of participants treated with the Connected Catheter with improved overall quality of life as measured by the SCI-QOL Survey and other surveys
UTI occurrence rate | 35-40 days
  Rate of participants treated with the Connected Catheter reported with a urinary tract infection
Lower Urinary Tract injury rate | 35-40 days
  Rate of participants treated with the Connected Catheter that experience a lower urinary tract injury

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - West Coast Urology, 11411 Brookshire Avenue, Suite 508, Downey, California
  - West Coast Urology, 575 E. Hardy St., Suite 215, Inglewood, California
  - Tri Valley Urology, 25495 Medical Center Dr., Suite 204, Murrieta, California
  - Chesapeake Urology, Owings Mills, Maryland
  - Minnesota Urology, 6025 Lake Road Suite 200, Woodbury, Minnesota
  - New Jersey Urology, 15000 Midlantic Drive, Suite 100, Mount Laurel, New Jersey
  - New Jersey Urology, 2401 Evesham Road, Suite F, Voorhees Township, New Jersey
  - Dr. Jonathan Vapnek Urology, New York, New York
  - Urology San Antonio, San Antonio, Texas